CLINICAL TRIAL: NCT04749264
Title: The Influence of Mindfulness Meditation Retreat on Attention to Internal Experience
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: TOVANA
Record Dates: First submitted 2020-12-20; First posted 2021-02-11 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2021-01

CONDITIONS: Attention Impaired; Cognitive Change; Mental Health Issue
Keywords: Internal attention; Interoceptive attention; Meditation; Mindfulness; Mindfulness Retreat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mindfulness Meditation Retreat: 6 to 7-days mindfulness meditation retreat
  Interventions: Behavioral: Mindfulness meditation retreat
- No intervention, Matched control: Adults participants will be recruited from social media and local community of meditation practitioners, and will be matched to the retreat group by gender, age and level of experience in meditation.

INTERVENTIONS:
Behavioral: Mindfulness meditation retreat — 6 to 7-days mindfulness retreat (Vipassana/insight meditation). The retreats are held in silence and led by senior teachers with many years of experience in teaching meditation. The focus of the retreat is the practice of mindfulness meditation while sitting and walking. Retreats include focused attention and open monitoring mindfulness meditation practices. Each retreat has a similar practice schedule thus the amount and nature of formal practice is mostly the same.
  Groups: Mindfulness Meditation Retreat

SUMMARY:
Although attention is thought to have a definitive functional role in mindfulness meditation training and its salutary mechanisms of action, extant empirical evidence is mixed and limited. In the proposed study, we propose to test whether 6 to 7-days mindfulness meditation retreats (N=90), relative to a wait-list control condition (N=45), will impact internal attentional processes or attention to internal experience (e.g., thoughts and bodily sensations); and whether these internal attentional change processes predict salutary outcomes of mindfulness meditation retreats. Participants will complete tasks designed to measure attention to internal experience before and then immediately following the retreat, as well as self-report measures of salutary outcomes before and 2-weeks post-retreat. Matched controls will complete the tasks at parallel time-points in the lab.

DETAILED DESCRIPTION:
Broadly, the investigators first aim is to assess whether mindfulness meditation retreat will yield significant improvement at post-relative to pre-retreat, compared to matched control, in each of these internal attentional processes: (i) enhanced ability to disengage from negative self-referential thoughts; (ii) reduced selection bias to negative self-referential thoughts; (iii) enhanced interoceptive attention and sensibility to a broader range of locations, intensities and hedonic tones of bodily sensations in response to negative and neutral self-referential thoughts; as well as (iv) enhanced mindful awareness during mindfulness meditation as expressed in the objects and temporal dynamics of mindful awareness. Second, the investigators will assess whether each of the aforementioned internal attentional change processes from pre- to post-retreat, will predict change from pre- to 2-weeks post-retreat in mindful awareness in daily living, mindfulness-related processes (e.g., decentering), and mental health. Third, investigators will assess whether previous meditation experience moderates these effects.

ELIGIBILITY:
Inclusion Criteria:

* Retreat Group: Adults who register to participate in a 6 to 7-days mindfulness meditation retreats.
* Control Group: Adults participants will be recruited from social media and local community of meditation practitioners, and will be matched to the retreat group by gender, age and level of experience in meditation.

Exclusion Criteria:

* Younger than 18 years-old and older than 65-years.
* Have first language other than Hebrew.
* Self-report lack of fluency in speaking or understanding Hebrew-language.
* Not having access to a computer and headphones with a microphone (for completing behavioral tasks).
* Participation in a retreat 1 month before the first primary outcomes assessment or during the weeks between the second primary outcomes assessment and the 2-weeks follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults from the general population and the local community of meditation practitioners.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Simulated Thought Paradigm - Digit Categorization Task | pre-intervention, immediately post-intervention
  The Simulated Thought Paradigm integrated into the Digit Categorization Task will be used to measure change, from pre-intervention to post-intervention, in internal attentional disengagement from simulated negative and neutral self-referential thoughts to a digit categorization (odd or even) task. Attentional disengagement will be computed via difference in reaction time to respond to digit target between negative and neutral self-referential thoughts. A positive score reflects greater difficulty to disengage from negative vs. neutral stimuli.
Change in Simulated Thought Paradigm - Dichotic 1-Back Task | pre-intervention, immediately post-intervention
  The Simulated Thought Paradigm integrated into the Dichotic 1-Back Task will be used to measure change, from pre-intervention to post-intervention, in internal selection between concurrent simulated negative and neutral self-referential thoughts. Biased selective internal attention will be computed via subtracting behavioral responding (e.g., accuracy) between concurrent negative and neutral self-referential thoughts. A positive bias score reflects greater selective attention to negative vs. neutral stimuli.
Change in Simulated Thought Paradigm - Body Map Task | pre-intervention, immediately post-intervention
  The Simulated Thought Paradigm integrated into the Body Map Task will be used to measure change, from pre-intervention to post-intervention, in interoceptive attention via subjective assessment (i.e. sensibility) of the frequency, location, intensity and hedonic tone of bodily sensations, as well as change in emotional experience (5-point Likert scale ranging from 1 to 5), in response to negative and neutral self-referential thoughts.
Change in Mindful Awareness Task | pre-intervention, 0-2 days post-intervention
  The Mindful Awareness Task is a behavioral paradigm will be used to measure change, from pre-intervention to post-intervention, in the objects and temporal dynamics of mindful awareness during mindfulness meditation. MAT scores include meta-awareness, quantified as the frequency of meta-awareness (i.e., awareness of the processes in consciousness); mindful awareness of body, mind, thoughts, pleasant and unpleasant hedonic tone, quantified as the frequency of mindful awareness of these experiential objects; mindful awareness time, quantified as the amount of time each participant engages in mindful awareness (in seconds); sustained mindful awareness, quantified as the average amount of time each participant sustains mindful-awareness without significant interruptions (in seconds); and latency to re-engagement in mindful awareness, quantified as the average amount of time it takes each participant to re-engage in mindful awareness following the onset of mindless states (in seconds).

SECONDARY OUTCOMES:
Change in Well-Being Index (WHO-5) | pre-intervention, 2-weeks post-intervention
  WHO-5 is a 5-item self-report questionnaire measuring well-being (6-point Likert scale ranging from 0 to 5) with higher scores indicating greater quality of life. The total score is the sum of all 5 items multiplied by 4 to create a score the ranges from 0 to 100. WHO will be used to measure change, from pre-to post-intervention, in well-being.
Change in Overall Anxiety Severity and Impairment Scale (OASIS) | pre-intervention, 2-weeks post-intervention
  OASIS is a 5-item self-report questionnaire measuring anxiety symptom severity (5-point Likert scale ranging from 0 to 4) with higher scores indicating greater anxiety-related severity and impairment. The total score is the sum of all 5 items, and ranges from 0 to 20. OASIS will be used to measure change, from pre-to post-intervention, in anxiety.
Change in Patient Health Questionnaire (PHQ-9) | pre-intervention, 2-weeks post-intervention
  PHQ-9 is a 9-item self-report questionnaire measuring depression symptom severity (4-point Likert scale ranging from 0 to 3) with higher scores indicating greater depression symptom severity. The total score is the sum of all 9 items, and ranges from 0 to 27. PHQ-9 will be used to measure change, from pre-to post-intervention, in depression.
Change in Perseverative Thinking Questionnaire (PTQ) | pre-intervention, 2-weeks post-intervention
  PTQ is a 15-items self-report questionnaire to measuring negative thinking that is repetitive, unproductive, difficult to disengage from and that captures mental capacity (5-point Likert-scale ranging from 0 to 4) with higher scores indicating greater repetitive thinking. The total score is the sum of all 15 items, and ranges from 0 to 60. PTQ will be used to measure change, from pre-to post-intervention, in negative repetitive thinking.
Change in Mind Wandering Questionnaire (MWQ) | pre-intervention, 2-weeks post-intervention
  MWQ is a 5-item self-report questionnaire measuring levels of mind-wandering (6-point Likert scale ranging from 1 to 6) with higher scores indicating greater levels of mind wandering. The total score is the sum of all 5 items, and ranges from 5 to 30. MWQ will be used to measure change, from pre-to post-intervention, in mind-wandering.
Change in Rumination Response Scale (RRS) - Brooding subscale | pre-intervention, 2-weeks post-intervention
  The brooding subscale of the RRS is a 5-items self-report questionnaire measuring levels of brooding (4-point Likert scale ranging from 1 to 4) with higher scores indicating greater levels of brooding. The total score is the sum of all 5 items, and ranges from 5 to 20. RRS will be used to measure change, from pre-to post-intervention, in rumination/brooding.
Change in The Five Facets Mindfulness Questionnaire (FFMQ) | pre-intervention, 2-weeks post-intervention
  FFMQ is a 39-item self-report questionnaire measuring 5 facets of trait mindfulness (5-point Likert scale ranging from 1 to 5) with higher scores indicating greater levels of trait mindfulness. The FFMQ includes 5 subscales measuring facets of mindfulness: observing, describing, acting with awareness, non-judging of experience, and non-reactivity to inner experience. Each subscale score is the sum of its items. FFMQ will be used to measure change, from pre-to post-intervention, in facets of trait mindfulness.
Change in The Multidimensional Assessment of Interoceptive Awareness (MAIA) | pre-intervention, 2-weeks post-intervention
  MAIA is a 32 -item self-report questionnaire measuring 8 dimensions of interoceptive awareness (6-point Likert scale ranging from 0 to 5) with higher scores indicating greater levels of interoceptive awareness. The MAIA includes 8 subscales measuring dimensions of interoceptive awareness: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Each subscale score is the sum of its items. MAIA will be used to measure change, from pre-to post-intervention, in dimensions of interoceptive awareness.
Change in Sussex-Oxford Compassion for the Self Scale (SOCS-S) | pre-intervention, 2-weeks post-intervention
  SOCS-S is a 20-item self-report questionnaire measuring 5 different dimensions of self-compassion (5-point Likert scale ranging from 1 to 5) with higher scores indicating greater levels of self-compassion. The SOCS-S includes 5 subscales measuring dimensions of self-compassion: recognizing suffering, understanding the universality of suffering, feeling for the person suffering, tolerating uncomfortable feelings, and motivation to act/acting to alleviate suffering. Each subscale score is the sum of its items. SOC-S will be used to measure change, from pre-to post-intervention, in dimensions of self-compassion.
Change in Metacognitive Processes of Decentering Scale - Trait (MPod-t) | pre-intervention, 2-weeks post-intervention
  MPod-t is a 15-item self-report questionnaire measuring trait levels of the 3 metacognitive processes of decentering (5-point Likert scale ranging from 1 to 5), with higher scores indicating greater levels of decentering. The MPoD-t includes 3 subscales measuring the metacognitive processes of decentering: meta-awareness, disidentification from internal experience, and non-reactivity to internal experience. Each subscale score is the sum of its items. MPod-t will be used to measure change, from pre-to post-intervention, in the metacognitive processes of decentering.
Change in The 7-Item Nonattachment Scale (NAS-7) | pre-intervention, 2-weeks post-intervention
  NAS-7 is a 7-item self-report questionnaire measuring nonattachment (6-point Likert scale ranging from 1 to 6) with higher scores indicating greater levels of nonattachment. The total score is the sum of all 7 items, and ranges from 7 to 42. NAS-7 will be used to measure change, from pre-to post-intervention, in nonattachment.
Change in The 16 item Difficulties in Emotion Regulation Scale (DERS-16) | pre-intervention, 2-weeks post-intervention
  DERS is a 16-item self-report questionnaire measuring 5 dimensions of difficulties in emotion regulation (5-point Likert scale ranging from 1 to 5) with higher scores indicating greater difficulties with emotion regulation. The DERS-16 includes 5 subscales measuring dimensions of difficulties in emotion regulation: lack of emotional clarity, difficulties engaging in goal-directed behavior, impulse control difficulties, limited access to effective emotion regulation strategies, nonacceptance of emotional responses. Each subscale score is the sum of its items. DERS-16 will be used to measure change, from pre-to post-intervention, in difficulties in emotion regulation.
Change in Trait International - Positive and Negative Affect Schedule - Short Form (I-PANAS-SF) | pre-intervention, 2-weeks post-intervention
  The trait I-PANAS-SF is a 10-item self-report questionnaire measuring trait positive and negative affect (5-point Likert scale ranging from 1 to 5) with higher scores indicating greater positive and negative affect. The I-PANAS-SF includes 2 subscales, one measuring positive affect and the other measuring negative affect. Each subscale score is the sum of its items. PANAS-SF will be used to measure change, from pre-to post-intervention, in negative and positive affect.
Change in State Mindfulness Scale (SMS) | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  SMS is a 21-item self-report questionnaire measuring state mindful awareness of body and mind (5-point Likert-type scale ranging from 1 to 5) during the MAT mindfulness meditation, with higher scores indicating greater state mindfulness. The SMS total score is the sum of all 21 items, and ranges from 21 to 105. It includes 2 subscales, one measuring mindful awareness of body and the other measuring mindful awareness of mind. Each subscale score is the sum of its items. SMS will be used to measure change, from pre-to post-intervention, in state mindfulness during the MAT mindfulness meditation.
Change in Toronto Mindfulness Scale - Curiosity subscale (TMS-C) | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  The curiosity subscale subscale of the TMS is a 6-item self-report questionnaire measuring state curiosity towards present moment experience (5-point Likert-type scale ranging from 0 to 4) during the MAT mindfulness meditation, with higher scores indicating greater state curiosity. The TMS-C score is the sum of all 6 items, and ranges from 0 to 24. TMS-C will be used to measure change, from pre-to post-intervention, in state curiosity during the MAT mindfulness meditation.
Change in Metacognitive Processes of Decentering Scale - State (MPod-s) | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  MPod-s is a 3-item self-report questionnaire measuring state levels of the 3 metacognitive processes of decentering (11-point Likert scale ranging from 0 to 10) with higher scores indicating greater levels of decentering (minimum scale score 0 and maximum scale score 10). Each of the 3 MPoD-s items measures a metacognitive process of decentering: meta-awareness, disidentification from internal experience, and non-reactivity to internal experience. MPod-s will be used to measure change, from pre-to post-intervention, in state decentering during the MAT mindfulness meditation.
Change in State International - Positive and Negative Affect Schedule - Short Form (State I-PANAS-SF) | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  State I-PANAS-SF is a 10-item self-report questionnaire measuring state positive and negative affect (5-point Likert scale ranging from 1 to 5) during the MAT mindfulness meditation, with higher scores indicating greater state positive and negative affect. The I-PANAS-SF includes 2 subscales, one measuring positive affect and the other measuring negative affect. Each subscale score is the sum of its items. State I-PANAS-SF will be used to measure change, from pre-to post-intervention, in state positive and negative affect during the MAT mindfulness meditation.
Change in Experience Sampling of Mindful Awareness During Meditation | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  11 experience sampling item measuring the following mindful awareness processes (9-point Likert scale ranging from 1 to 9) during the MAT mindfulness meditation: mindful awareness of the breath, body, mind, pleasant and unpleasant hedonic tone, as well as meta-awareness, mindful awareness time, sustained mindful awareness, and latency to re-engagement in mindful awareness, and mindful awareness of change. Higher scores indicate greater levels of mindful awareness. Experience sampling will be used to measure change, from pre-to post-intervention, in state mindful awareness processes during the MAT mindfulness meditation.
Change in Experience Sampling of Attitudinal Qualities of Mindfulness During Meditation | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  9 experience sampling item measuring the following attitudinal qualities of mindful awareness (9-point Likert scale ranging from 1 to 9) during the MAT mindfulness meditation: curiosity about bodily and mental experience, distance and (dis)Identification with internal experience, hedonic-based desire of pleasant and unpleasant experience (non-equanimity), willingness, and experiential avoidance. Higher scores indicate greater levels of each attitudinal quality. Experience sampling will be used to measure change, from pre-to post-intervention, in attitudinal qualities of mindful awareness during the MAT mindfulness meditation.
Change in Experience Sampling of Phenomenological States During Meditation | immediately after MAT administration pre-intervention, immediately after MAT administration post-intervention
  9 experience sampling item measuring the following phenomenological states (9-point Likert scale ranging from 1 to 9) during the MAT mindfulness meditation: fatigue, alertness, falling asleep, effort, boredom, enjoyment, relaxation, and mind-wandering frequency and duration. Higher scores indicate greater levels of each phenomenological state. Experience sampling will be used to measure change, from pre-to post-intervention, in phenomenological states during the MAT mindfulness meditation.
Peak Meditative Experience Scale (PMES) | 0-2 days post-intervention
  PMES is a 32-item self-report questionnaire measuring the occurrence of 32 types of peak experiences (unusual and uncommon experiences) during the retreat/last week ("yes" or "no"), their frequencies (open ended number), duration (open ended number), and degree of hedonic tone (9-point Likert scale ranging from -4 to +4). Positive hedonic tone scores indicate pleasant hedonic tone, zero scores indicate neutral hedonic tone, negative scores indicate unpleasant hedonic tone. The PMES items relate to 6 domains of peak experiences: positive emotions, negative emotions, perception, altered states of consciousness, dissociation, and insight.
Impact of Peak Meditative Experience Scale (I-PMES) | 2-weeks post-intervention
  I-PMES is a self-report questionnaire measuring the positive and negative impact of peak experiences that participants had during the retreat, on participant's lives after the retreat (two 5-point Likert scales for each experience: positive impact ranging from 0 to +4, negative impact ranging from 0 to -4). The number of items in this scale varies between participants as they are only asked to rate the impact of peak experiences they indicated in the PMES that they had during the retreat. Only participants in the mindfulness meditation retreat condition will complete this measure.

OTHER OUTCOMES:
Previous Meditation Experience Interview | pre-intervention
  A structured phone interview assessing previous experience in meditation retreats and previous regular meditation practice. During this interview, participants are asked to specify each meditation retreat in which they participated in the past, and their previous regular meditation practice. The following scores are computed based on participants' reports: total number of days in mindfulness meditation retreats and total number of months and hours of previous regular mindfulness meditation practice outside of retreats (at least once a week). Similar scores are computed for previous retreats and regular practice of meditation styles that do not emphasize the cultivation of mindfulness (e.g., transcendental meditation).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bernstein, Ph.D., Principal Investigator — University of Haifa
Locations (1):
- Amutat Tovana, Afula, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Hadash Y, Veksler T, Dar O, Oren-Schwartz R, Bernstein A. Peak experiences during insight mindfulness meditation retreats and their salutary and adverse impact: A prospective matched-controlled intervention study. J Consult Clin Psychol. 2024 Apr;92(4):213-225. doi: 10.1037/ccp0000875. PMID 38573713